CLINICAL TRIAL: NCT05128994
Title: Keep it Simple: A Broadly Usable, High-performance Grasp Orthotic
Brief Title: Hand Grasp Function After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Battelle Memorial Institute (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 100144033
Record Dates: First submitted 2021-10-19; First posted 2021-11-22 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; functional electrical stimulation; hand function
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Non-invasive FES (Experimental): Wearable FES sleeve with non-invasive user controls
  Interventions: Device: User-controlled FES system

INTERVENTIONS:
Device: User-controlled FES system — Wearable FES sleeve with non-invasive user controls

SUMMARY:
The objective of this study is to advance personalized, portable, and non-invasive hand-grasp neuro-orthoses that restore naturalistic grasp functions for those with tetraplegia due to spinal cord injury (SCI), designed around their needs and preferences.

DETAILED DESCRIPTION:
Battelle has developed a novel wearable sleeve that can reanimate a paralyzed limb via Functional Electrical Stimulation (FES) that is controlled non-invasively by the user. Previous work has shown the ability of this sleeve and FES technology to significantly enhance independence and quality of life when controlled by an implanted brain-computer interface, thus now investigators plan to trial use of the high-definition FES system with simpler, non-invasive control mechanisms to expedite translation of this technology into real-world settings. Each participant will complete up to 10 research sessions (~1.5hrs each) in their residence or at an alternative location. The study location is restricted to Columbus Ohio and surrounding areas. Participants will be compensated for their time.

In Aim 1, investigators will evaluate the ability of a non-invasive, user-controlled FES system to increase functional hand use in the homes of individuals with SCI. The research team will train participants to use the FES system for different functional hand movements and activities they identify as important to them, then measure FES system effectiveness using standardized assessments.

In Aim 2, investigators will assess the viability of using the sleeve technology to non-invasively record muscle activity as the participant attempts different functional movements.

In Aim 3, human-centric design methodology and contextual inquiry interviews will be employed to understand study participants' needs and preferences for a FES assistive device. This information will determine actions to improve usability and optimize the system for unsupervised home use.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* ≥ 12 months post-SCI and medically/neurologically stable
* Cervical spinal cord injury (C1-C8); any etiology except neurodegenerative conditions
* Unable to grasp objects independently with both hands (tetraplegia)
* Manual muscle testing (MMT) scores ≥4/5 for elbow flexion and ≥2/5 for wrist extension
* Willing to participate in sessions at home or able to travel to alternate site for study sessions

Exclusion Criteria:

* Ventilator-dependent (dependent upon mechanical life support due to inability to breathe effectively)
* Poorly controlled autonomic dysreflexia (more than one episode in 3 months prior to enrollment)
* Moderate to severe spasticity (Modified Ashworth Scale (MAS) >1+) in the hand, wrist, or forearm
* Received a localized injection (e.g. Botox) to hand, wrist, or forearm muscles within past 12 months
* Currently participating in physical rehabilitation for upper extremity impairments
* Individuals having or requiring any of the following: implanted pacemaker, life supporting/sustaining equipment, or critical non-removable implantable electronic devices such as an insulin pump or neurostimulator.
* Presence of any other clinically significant medical comorbidity and/or neurological condition for which participation in the study may pose a safety risk and/or influence results
* Presence of the following medical conditions: uncontrolled seizure disorder, active malignancy in the upper extremities, or open wounds/infections in the upper extremities
* Individuals whose forearm is determined to be too small or too large to fit the electrode sleeve being investigated
* Individuals who are pregnant or plan to get pregnant during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of FES sleeve as a functional orthosis for activities of daily living | 10 weeks
  Semi structured interviews will involve gaining participants opinions on the strengths and weaknesses of the system

SECONDARY OUTCOMES:
Quadriplegia Index of Function (QIF) | At study completion, 10 weeks
  Self-report tool assessing 37 activities of daily living with each task scored from 0 to 4 in order of increasing independence.
Change in Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) after 10 weeks | 10 weeks
  Standardized test will assess participant's ability to perform complex grasp tasks: pouring a bottle; opening lids on two sizes of jars; inserting/turning key in lock; manipulating pegs in a pegboard; inserting four sizes of coins into slots; and screwing four sizes of nuts onto bolts
Psychosocial Impact of Assistive Devices Scale (PIADS) | At study completion, 10 weeks
  Assesses user opinions of assistive devices across 26 items, describing likelihood of device adoption for regular use and psychosocial effects of use on function independence, well-being, and quality of life. Each item is scored on a 7 point Likert Scale from -3 to 3 with higher scores indicating more positive impact.
Change in Electromyography (EMG) signal metrics | 10 weeks
  Metrics derived from noninvasively recorded electromyography activity as the user attempts functional hand movements
Number of serious adverse events | 10 weeks
  Assessed by number of incidences

OTHER OUTCOMES:
Setup time (minutes) | 10 Weeks
  The time it takes to physically don, connect, and calibrate system components
Canadian Occupational Performance Measure (COPM) | Week 1, First session
  A 9 item assessment to measure perceived occupational performance of self-care, productivity and leisure. COPM uses semi-structured interview questions to identify activities that the individuals wants, needs or is expected to perform.

CONTACTS AND LOCATIONS:
Overall Officials: David A Friedenberg, PhD, Principal Investigator — Battelle
Locations (1):
- Battelle Memorial Institute, Columbus, Ohio, United States